CLINICAL TRIAL: NCT05993182
Title: Comparative Study Among Different Doses of Ephedrine During Elective Cesarean Section Under Subarachnoid Block - Time to Event Analysis.
Brief Title: Comparative Study Among Different Doses of Ephedrine During Elective Cesarean Section Under Subarachnoid Block.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Ayman Mohamady Eldemrdash, Doctor Ayman Mohamady Eldemrdash, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 669/10/22
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; Cesarean Section Complications; Subarachnoid Block
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-I (Active Comparator): received 5mg of Ephedrine after the first hypotension [ Base line time or starting point is first hypotension]
  Interventions: Drug: Ephedrine 5mg
- Group-II (Active Comparator): received 10mg of Ephedrine after the first hypotension [ Base line time or starting point is first hypotension]
  Interventions: Drug: Ephedrine 10mg
- Group-III (Active Comparator): 15mg bolus dose of ephedrine IV after the first hypotension [ Base line time or starting point is first hypotension]
  Interventions: Drug: Ephedrine 15mg

INTERVENTIONS:
Drug: Ephedrine 5mg — Patients received 5mg bolus dose of ephedrine Intravenous after the first hypotension [ Base line time or starting point is first hypotension]
  Arms: Group-I
Drug: Ephedrine 10mg — Patients received 10mg bolus dose of ephedrine Intravenous after the first hypotension [ Base line time or starting point is first hypotension]
  Arms: Group-II
Drug: Ephedrine 15mg — Patients received 15mg bolus dose of ephedrine Intravenous after the first hypotension [ Base line time or starting point is first hypotension]
  Arms: Group-III

SUMMARY:
compare the time of second hypotension after administration of three different doses of ephedrine 5,10,15 mg

DETAILED DESCRIPTION:
In cesarean section, under subarachnoid block the most common complication is hypotension with a reported incidence greater than 80%. Hypotension may occur even after left uterine displacement and preloading with crystalloid. The severity of hypotension depends on the degree of aortocaval compression syndrome, the amount of crystalloid preloading, doses of local anesthetic drugs administered. The most effective treatment of hypotension associated with cesarean section under subarachnoid block is the administration of vasopressor drugs.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists 1 and 2 patients
* Gestational amenorrhea of > 32 weeks
* Elective cesarean section
* Patient willing for spinal anesthesia.
* Singleton pregnancy with cephalic presentation.
* Baseline systolic blood pressure between 100-140 mmHg and diastolic blood pressure between 70-89 mmHg.

Exclusion Criteria:

* Any contraindication to spinal anesthesia, i.e., local infection at the site of injection
* valvular heat diseases
* bleeding tendency
* any co-morbidity like diabetes mellitus
* liver cirrhosis
* renal failure
* any obstetric complications like placenta previa
* pregnancy-induced hypertension or HELLP syndrome
* multiple gestations
* fetal malformation
* coagulopathies
* morbid obesity and spine deformity
* profound hypotension (total spinal) bradycardia and need atropine and severe bleeding

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Survival analysis or time until an event occurs | Intraoperatively
  The study time is a30 minute and blood pressure is measured automatically non invasive at 3-minute intervals. If systolic blood pressure decreased more than 20% from the baseline(Event)

SECONDARY OUTCOMES:
Starting point or Base line time | Intraoperatively
  Starting point or Base line time is a first hypotension
Survival time | Intraoperatively
  Free of event(No hypotension) at any time after base line

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author